CLINICAL TRIAL: NCT02590016
Title: Glucose Control During Labour in Gestational Diabetes Mellitus With Insulin Treatment: Insulin-Glucose-Infusion Versus Observational Approach - Is There a Difference in Neonatal Hypoglycemia Rate?
Brief Title: Glucose Control During Labour in Gestational Diabetes Mellitus With Insulin Treatment: A Randomized Controlled Trial
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tampere University Hospital (Other)
Responsible Party: Principal Investigator, Elina Kivekäs, MD, Tampere University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R15050M
Record Dates: First submitted 2015-10-21; First posted 2015-10-28 (Estimated); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: Gestational Diabetes; Hypoglycemia, Neonatal
MeSH Terms: conditions — Diabetes, Gestational; Hypoglycemia | interventions — Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Insulin-glucose-infusion (Experimental): Insulin-glucose-infusion is administered once active labour begins and will be continued until birth.
  Interventions: Drug: Insulin, Aspart
- Observation (Active Comparator): Plasma glucose level is measured every 1-2 hours during active labour and insulin-glucose-infusion is started if plasma glucose level exceeds 7,5 mmol/l in two subsequent measurements.
  Interventions: Drug: Insulin, Aspart

INTERVENTIONS:
Drug: Insulin, Aspart — Insulin aspart Novorapid® Penfill 40 IU/0,4 ml is diluted into 1000ml of 0,9 % sodium chloride (NaCl). Infusion is started at rate 48 ml/l, which equates insulin dosing at rate of 2 IU/h. Glucose infusion is started simultaneously. 5 ml of potassium chloride (KCl) is added to 500 ml of 10 % Glucose solution. Infusion rate is 100 ml/h giving glucose infusion rate of 10 g/l. Plasma glucose level is measured every 1-2 hours and infusion rate of insulin is increased by 6ml/h if plasma glucose is more than 7,5 mmol/l and decreased by 6 mmol/h if plasma glucose is below 4 mmol/l.
  Other Names: Novorapid

SUMMARY:
Pregnant women with gestational diabetes who are treated with insulin and their daily insulin dose is 30 IU or more will be randomized into two groups. Active treatment group will receive insulin-glucose-infusion during labour. In the observational group, blood glucose level during labour will be monitored and insulin-glucose-infusion is started only if needed. The hypothesis is that there will not be a difference in rate of hypoglycemia between the two groups and that the proportion of observational group participants that need infusion is low.

DETAILED DESCRIPTION:
Intrapartum blood glucose level has negative correlation to neonatal blood glucose level in type 1 diabetics. In gestational diabetes the correlation is less clear. In the view of current knowledge, it seems that moderately elevated intrapartum blood glucose may not cause neonatal hypoglycemia. There is no consensus of how to treat intrapartum blood glucose level in gestational diabetics. Some studies have implied that most of mothers with gestational diabetes would have normal blood glucose level during labour and hence would not need any intervention if their daily insulin dosage is less than 0,5-1 IU/kg.

Study participants are recruited into the study at Tampere University Hospital Maternity Ward when their daily insulin dose exceeds 30 IU. Randomization is done at 37th gestational week, if vaginal delivery is planned, and HbA1c is measured. Randomization envelope is opened at the delivery ward when active labour begins and treatment of blood glucose level is carried out accordingly. If insulin dose is 1 IU/kg or more, the participant is treated as in active treatment group despite of result of randomization. All neonates will receive milk substitute after birth in labour ward. Plasma glucose is measured immediately if neonate has symptoms of low blood sugar. If not, plasma glucose is measured approximately two hours after birth and after that every 4 hours until plasma glucose is 3,0 mmol/l or more in three consecutive measurements.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women with gestational diabetes mellitus and daily insulin dosage of 30 IU or more

Exclusion Criteria:

* planned caesarean section,
* premature birth (< 37 gestational weeks)

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-09; Primary Completion 2020-12 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Neonatal hypoglycemia | within 48 hours after birth
  Neonatal plasma blood glucose < 3 mmol/l

SECONDARY OUTCOMES:
Moderate neonatal hypoglycemia | within 48 hours after birth
  Neonatal plasma blood glucose < 2,6 mmol/l
Severe neonatal hypoglycemia | within 48 hours after birth
  Neonatal plasma blood glucose <2,2 mmol/l and/or demand of treatment
Duration of neonatal blood glucose monitoring | within a week after birth
Proportion of participants needing insulin-glucose-infusion in the observational arm | during active labour

CONTACTS AND LOCATIONS:
Overall Officials: Elina Kivekäs, MD, Principal Investigator — Obstetrics and Gynecology Unit: Tampere University Hospital
Locations (1):
- Obstetrics and Gynecology Unit: Tampere University Hospital, Tampere, Finland

REFERENCES:
- [Background] Barrett HL, Morris J, McElduff A. Watchful waiting: a management protocol for maternal glycaemia in the peripartum period. Aust N Z J Obstet Gynaecol. 2009 Apr;49(2):162-7. doi: 10.1111/j.1479-828X.2009.00969.x. PMID 19432604
- [Background] Flores-le Roux JA, Sagarra E, Benaiges D, Hernandez-Rivas E, Chillaron JJ, Puig de Dou J, Mur A, Lopez-Vilchez MA, Pedro-Botet J. A prospective evaluation of neonatal hypoglycaemia in infants of women with gestational diabetes mellitus. Diabetes Res Clin Pract. 2012 Aug;97(2):217-22. doi: 10.1016/j.diabres.2012.03.011. Epub 2012 Apr 24. PMID 22537519
- [Background] Garabedian C, Deruelle P. Delivery (timing, route, peripartum glycemic control) in women with gestational diabetes mellitus. Diabetes Metab. 2010 Dec;36(6 Pt 2):515-21. doi: 10.1016/j.diabet.2010.11.005. PMID 21163417
- [Background] Maayan-Metzger A, Lubin D, Kuint J. Hypoglycemia rates in the first days of life among term infants born to diabetic mothers. Neonatology. 2009;96(2):80-5. doi: 10.1159/000203337. Epub 2009 Feb 19. PMID 19225239
- [Background] Metzger BE, Persson B, Lowe LP, Dyer AR, Cruickshank JK, Deerochanawong C, Halliday HL, Hennis AJ, Liley H, Ng PC, Coustan DR, Hadden DR, Hod M, Oats JJ, Trimble ER; HAPO Study Cooperative Research Group. Hyperglycemia and adverse pregnancy outcome study: neonatal glycemia. Pediatrics. 2010 Dec;126(6):e1545-52. doi: 10.1542/peds.2009-2257. Epub 2010 Nov 15. PMID 21078733
- [Background] Stenninger E, Schollin J, Aman J. Early postnatal hypoglycaemia in newborn infants of diabetic mothers. Acta Paediatr. 1997 Dec;86(12):1374-6. doi: 10.1111/j.1651-2227.1997.tb14916.x. PMID 9475319
- [Background] Ryan EA, Al-Agha R. Glucose control during labor and delivery. Curr Diab Rep. 2014 Jan;14(1):450. doi: 10.1007/s11892-013-0450-4. PMID 24292970
- [Background] Ryan EA, Sia WW, Khurana R, Marnoch CA, Nerenberg KA, Ghosh M. Glucose control during labour in diabetic women. J Obstet Gynaecol Can. 2012 Dec;34(12):1149-1157. doi: 10.1016/S1701-2163(16)35462-7. PMID 23231797